CLINICAL TRIAL: NCT04358510
Title: Mortality Prediction Model for the Triage of COVID-19, Pneumonia and Mechanically Ventilated ICU Patients
Brief Title: COVID-19 Mortality Prediction Model
Status: Completed | Type: Observational
Sponsor: Dascena (Industry)
Responsible Party: Sponsor
Other Study IDs: 04202001
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; Pneumonia; Mechanical Ventilation
Keywords: machine learning; COVID-19; mortality; prediction; pneumonia; mechanical ventilation
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COViage: Machine learning intervention
  Interventions: Device: COViage

INTERVENTIONS:
Device: COViage — The COViage machine learning algorithm is designed to predict mortality in COVID-19, pneumonia and mechanically ventilated ICU patients.

SUMMARY:
The objective of this study is to develop and evaluate an algorithm which accurately predicts mortality in COVID-19, pneumonia and mechanically ventilated ICU patients.

DETAILED DESCRIPTION:
Retrospective study of 53,001 total ICU patients, including 9,166 patients with pneumonia and 25,895 mechanically ventilated patients, performed on the MIMIC dataset. The NPH patient dataset includes 114 patients positive for SARS-COV-2 by PCR test.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Record of ICU stay

Exclusion Criteria:

* Patients aged less than 18 years
* Patients for which there were no records of raw data or no discharge or death dates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective study of 53,001 total ICU patients, including 9,166 patients with pneumonia and 25,895 mechanically ventilated patients, performed on the MIMIC dataset. The community hospital patient dataset included 114 patients positive for SARS-COV-2 by PCR test.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Mortality outcome in COVID-19 ICU patients | Through study completion, an average of 2 months
  Deceased or not deceased
Mortality outcome in mechanically ventilated ICU patients | Through study completion, an average of 2 months
  Deceased or not deceased
Mortality outcome in pneumonia ICU patients | Through study completion, an average of 2 months
  Deceased or not deceased

CONTACTS AND LOCATIONS:
Locations (1):
- Dascena, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: Undecided